CLINICAL TRIAL: NCT06344936
Title: Open-Label Assessment of the Effects of Itraconazole and Rifampicin on HRS-1780 Pharmacokinetics in Healthy Subjects
Brief Title: Drug-drug Interaction Study of HRS-1780 Tablets in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1780-103
Record Dates: First submitted 2024-03-22; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease(CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental)
  Interventions: Drug: HRS-1780 tablets; Itraconazole capsules; Rifampicin capsules

INTERVENTIONS:
Drug: HRS-1780 tablets; Itraconazole capsules; Rifampicin capsules — Treatment PartⅠ: Itraconazole capsule, 200mg QD, 7 times; HRS-1780 tablets, 10mg QD, twice Treatment PartⅡ: Rifampicin capsules, 600mg QD, 14 times; HRS-1780 tablets, 10mg QD, twice

SUMMARY:
The study was designed to evaluate the pharmacokinetic effects of itraconazole and rifampicin on HRS-1780 after oral administration of HRS-1780 tablets in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent before the test, fully understand the test content, process and possible adverse reactions, and be willing to complete the study according to the requirements of the test plan;
2. Healthy participants aged 18 to 45 years old (including both ends) on the date of signing the informed consent;
3. Male participants weigh no less than 50kg, female participants weigh no less than 45kg, and body mass index (BMI) is in the range of 19.0~26.0 kg/m2 (including the cut-off value).
4. The participant (including the partner) does not have a family plan and voluntarily takes the contraceptive measures specified in the program within 3 months after signing the informed consent letter to the last medication; Participants did not plan to donate sperm or eggs within 3 months after the end of the last dose.

Exclusion Criteria:

1. Those who participated in blood donation and donated ≥400mL of blood within 3 months before taking the study drug, or received blood transfusion;
2. Allergic constitution, including allergy related diseases (eczema, urticaria, allergic rhinitis, etc.), drug allergy or drug allergic reaction history; History of allergy to HRS-1780 tablets, itraconazole, rifampicin, rifamycin or its excipients;
3. Have a history of drug and/or alcohol abuse, test positive for alcohol and drugs or have a history of drug abuse in the past five years or use of drugs in the three months prior to the test;
4. Drinking more than 14 units of alcohol per week in the 6 months prior to screening (1 unit = 285mL for beer, 25mL for spirits, or 100mL for wine); Or have taken alcohol-containing products 48 hours before administration; Or positive alcohol breath test at baseline. ;
5. Smoking more than 5 cigarettes per day in the 3 months before screening or use of any tobacco products 48 hours before dosing.
6. Patients with abnormal vital signs, comprehensive physical examination, routine laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function), 12-lead electrocardiogram, chest X-ray, abdominal B-ultrasonography and judged by the investigator to be clinically significant;
7. Medical history of major organ diseases, such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and skeletal musculoskeletal system, is not considered suitable for participation in this study;
8. Patients with severe systemic infectious diseases, severe trauma or major surgical operations in the 3 months prior to screening and who plan to undergo surgery during the trial;
9. Have participated in a clinical trial of any drug or medical device within 3 months or 5 half-lives prior to screening, whichever is longer, or plan to participate in a clinical trial of another drug or medical device during the trial period;
10. Have taken any prescription or over-the-counter drugs in the 14 days prior to taking the study drug;
11. HCV antibody positive, HIV antibody positive, HBsAg positive, syphilis antibody positive;
12. Women of childbearing age who have positive blood pregnancy tests at baseline;
13. Pregnant and lactating women;
14. Patients with a history of needle fainting and blood fainting, difficulty in blood collection or inability to tolerate venous puncture blood collection;
15. Those who could not follow the dietary requirements during the trial;
16. Subjects with other factors deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Assess the Cmax of HRS-1780 in plasma. | About 3 days after the dose.
Assess the Tmax of HRS-1780 in plasma. | About 3 days after the dose.
Assess the t1/2 of HRS-1780 in plasma. | About 3 days after the dose.
Assess the AUC0-t of HRS-1780 in plasma. | About 3 days after the dose.
Assess the AUC0-inf of HRS-1780 in plasma. | About 3 days after the dose.

SECONDARY OUTCOMES:
Assess the incidence and severity of adverse events in healthy subjects after administration of HRS-1780 tablets. | About a month from the first medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided